CLINICAL TRIAL: NCT06939816
Title: A Study to Assess the Effect of Vonafexor on Kidney Function in Subjects With Impaired Renal Function and Suspected MASH
Brief Title: Vonafexor in Patients With Impaired Renal Function and Suspected MASH (Metabolic Dysfunction-associated Steatohepatitis)
Acronym: MASH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EYP001-210; 2023-509192-16-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease Stage 2; Chronic Kidney Disease Stage 3; Metabolic Dysfunction-Associated Steatohepatitis
Keywords: CKD; Chronic Kidney Disease; MASH; Metabolic Dysfunction-Associated Steatohepatitis; Kidney function; eGFR; estimated Glomerular function rate; mGFR; measured Glomerular function rate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vonafexor low dose (Experimental): Vonafexor low dose 1 tablet per day
  Interventions: Drug: Vonafexor low dose
- Vonafexor high dose (Experimental): Vonafexor high dose 1 tablet per day
  Interventions: Drug: Vonafexor high dose

INTERVENTIONS:
Drug: Vonafexor low dose — Oral tablets
  Arms: Vonafexor low dose
Drug: Vonafexor high dose — Oral tablets
  Arms: Vonafexor high dose

SUMMARY:
This study is designed to establish the effect of 2 doses of vonafexor on the kidney. This will be investigated in subjects with mild or moderate reduced estimated glomerular filtration rate (eGFR) and suspected MASH. In addition, the non-invasive multiparametric magnetic resonance imaging assessment of functional and structural changes in the kidney and in the liver will be investigated.

DETAILED DESCRIPTION:
This is a phase 2, open-label, two-dose, randomized, parallel arms, single center study where subjects are participating for up to 32 weeks:

* Screening: 4 weeks
* Treatment: 16 weeks
* Follow-up: 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before any trial-related activities
* Male or female subject.
* Age between 18 and 75 years, both inclusive.
* Overweight or obesity (body mass index BMI ≥ 25.0 kg/m2 and ≤ 45.0 kg/m2) with or without type 2 diabetes mellitus (T2DM with an HbA1c ≤ 9.5%).
* eGFR ≥ 30 and < 90 (mL/min/1.73 m²).
* Presumed mild to higher liver fibrosis as shown by a FIBROTEST score ≥ 0.28 and/or FIB-4 score ≥ 1.3.

Exclusion Criteria:

* Known or suspected hypersensitivity to IMP or any of the excipients or to any component of the IMP formulation.
* Previous participation in this trial. Participation is defined as randomised.
* Receipt of any medicinal product in clinical development within 30 days or at least 5 half-lives of the related substances and their metabolites (whichever is longer) before randomisation in this trial.
* History of multiple and/or severe allergies to drugs including contrast media or foods or a history of severe anaphylactic reaction.
* Known non-MASH liver disease.
* History or presence of cirrhosis (evidenced on imaging or by histology, or liver decompensation, including ascites, hepatic encephalopathy, or presence of esophageal varices).
* Total body weight loss of >5% within 6 months prior to screening.
* If female, pregnancy or breast-feeding.
* Women of childbearing potential who are not using a highly effective contraceptive method and whose male partner is not using a highly effective contraceptive method for the entire study duration and for at least 6 weeks after last dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of mGFRiohexol at week 16 | 16 weeks
Change from baseline of eGFRcreatinine at week 16 | 16 weeks

SECONDARY OUTCOMES:
Vonafexor plasma concentrations | 16 weeks
  Plasma concentrations pre-dose and post-dose which will be modelled against the MASH PopPK expected values
Change from baseline mGFRiohexol off treatment at week 24 | 24 weeks
Change from baseline of eGFRcreatinine on treatment at weeks 4, 8, 12 and off treatment at weeks 20, 24 and 28 | 28 weeks
Correlation of mGFRiohexol with eGFRcreatinine at baseline, on treatment at week 16 and off treatment at week 24 | 24 weeks
Levels and change in proteinuria in morning urine samples at baseline, on treatment at weeks 4, 8, 12, 16 with off treatment at weeks 20, 24 and 28 | 28 weeks
Treatment-emergent adverse events and serious adverse events | 28 weeks

OTHER OUTCOMES:
MRI kidney biomarkers time course from baseline, to on treatment at week 16 and to off treatment at week 24 | 24 weeks
MRI liver biomarkers time course from baseline, to on treatment at week 16 and to off treatment at week 24 | 24 weeks
Liver biomarker FIB-4 changes from baseline at on treatment week 8, 16 and off treatment at week 24 | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline published results might be shared upon request with researchers who provide a methodologically sound proposal and to achieve objectives as set in the approved proposal.
  IPD will be shared deidentified and from 3 months and ending 5 years following article publication.